CLINICAL TRIAL: NCT05717270
Title: Two-layer Suturing of Achilles Tendon Ruptures - an Ambidirectional Cohort Study
Brief Title: Two-layer Suturing of Achilles Tendon Ruptures
Acronym: ATRBFH
Status: Active, not recruiting | Type: Observational
Sponsor: Bispebjerg Hospital (Other)
Responsible Party: Principal Investigator, Anne-Sofie Agergaard, Project administrator, Bispebjerg Hospital
Other Study IDs: ATR_sutur_BFH
Record Dates: First submitted 2023-01-26; First posted 2023-02-08 (Actual); Last update posted 2024-09-27 (Actual); Status verified 2024-09

CONDITIONS: Achilles Tendon Rupture

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Patient Registry: Yes
Target Follow-Up Duration: 12 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Prospective group: Acute Achilles tendon Rupture undergoing surgical repair.
  Interventions: Procedure: Two-layered suture repair
- comparison group: Patients group from a previous trial (NCT04263493).

INTERVENTIONS:
Procedure: Two-layered suture repair — The ruptured Achilles tendon will be sutured in two-layer.
  Groups: Prospective group

SUMMARY:
The purpose of the present study is to measure whether a new technique of double row suturing of a ruptured Achilles tendon will result in a normalization of the length of the Soleus part (primary outcome) and of the superficial Gastrocnemius part of the tendon (secondary outcome) one-week post-operative. Results will be compared to that of a participants group that underwent the same operation but with a standard operative technique and the same rehabilitation regime recently completed (NCT04263493).

The investigators hypothesize that the new suturing technique will result in an elongation of the Soleus part of the Achilles tendon (primary outcome) by 8.9 mm or less relative to the uninjured contralateral side one week (primary endpoint) after surgery compared to retrospective data from a recently completed randomized controlled trial

DETAILED DESCRIPTION:
This study is an ambidirectional cohort study with a retrospective part based on a recently completed trial (NCT04263493) and this prospective registered trial.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed with a traumatic, complete mid-substance Achilles tendon rupture
* Manages transportation to/from the hospital on their own
* Presented within 14 days from injury
* Adult (18 to 60 years)
* Understands Danish

Exclusion Criteria:

* Other injuries affecting their lower limb functions
* Prior Achilles contralateral tendon rupture
* Contraindications for MRI
* Re-rupture
* Smoking
* Systemic diseases influencing tendon healing
* Anticoagulation treatment
* Inability to follow rehabilitation or complete follow-ups
* Immunosuppressive treatment including systemic corticosteroid treatment.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: Patients with diagnosed acute Achilles tendon rupture
Sampling Method: Probability Sample
Enrollment: 23 (Estimated)
Dates: Start 2023-05-23 (Actual); Primary Completion 2025-02-01 (Estimated); Study Completion 2026-02-01 (Estimated)

PRIMARY OUTCOMES:
Tendon length | One week after surgery.
  The distance between the distal muscle fibers of the Soleus muscle and the posterior most superior part of the calcaneus.

SECONDARY OUTCOMES:
Tendon length Soleus | One week after surgery.
  The distance (mm) between the distal muscle fibers of the gastrocnemius muscle and the posterior most superior part of the calcaneus.
Tendon length Triceps Surae | 6 months.
  The soleus and gastrocnemius tendon length (mm).
Plantar flexion function | 6 and 12 months.
  Heel-rise test
Patient perception | 12 months
  Achilles Tendon Total Rupture Score (ATRS). The ATRS consist of 10 items, with a total score range from 0 to 100, and a low score indicate more limitations in physical activity and worse symptoms.
Vascularisation | 6 months.
  Doppler flow (area in mm2)
Muscle architecture fascicle length | 6 months.
  Gastrocnemius and soleus muscle fascicle length (mm).
Muscle architecture pennation angle | 6 months.
  Gastrocnemius and soleus muscle pennation angle (°).
Muscle cross sectional area | 6 months.
  Gastrocnemius and soleus tendon and lower limb muscle cross-sectional area (mm2).

CONTACTS AND LOCATIONS:
Locations (1):
- Institute of Sports Medicine Copenhagen, Copenhagen, NV, Denmark

IPD SHARING:
Plan to Share IPD: No